CLINICAL TRIAL: NCT02334748
Title: A French Open-label Extension Study of Canakinumab in Patients Who Participated in International Phase III Studies CACZ885G2301E1 or CACZ885G2306 in Systemic Juvenile Idiopathic Arthritis and CACZ885N2301 in Hereditary Periodic Fevers (TRAPS, HIDS, or crFMF)
Brief Title: A Study of Canakinumab in Patients With Systemic Juvenile Idiopathic Arthritis or Hereditary Periodic Fevers Who Participated in the CACZ885G2301E1, CACZ885G2306 or CACZ885N2301 Studies
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CACZ885GFR01; 2014-002872-95 (EudraCT Number)
Record Dates: First submitted 2014-12-23; First posted 2015-01-08 (Estimated); Results first posted 2020-05-19 (Actual); Last update posted 2020-05-19 (Actual); Status verified 2020-05

CONDITIONS: Systemic Juvenile Idiopathic Arthritis; Hereditary Periodic Fevers
Keywords: Juvenile Rheumatoid arthritis (JRA) chronic; systemic inflammatory disorder; painful joints; inflammation of the synovial membrane; auto-immune rheumatoid disease; reactive rheumatoid arthritis; Systemic Juvenile Rheumatoid arthritis (SJRA); Hereditary Periodic Fevers; Hereditary periodic fever syndrome(HPFS); Familial Mediterranean fever syndrome(FMFS); Hyperimmunoglobulinemia D; Tumor necrosis factor (TNF) receptor-associated periodic syndrome (TRAPS); Muckle-Wells syndrome (MWS); Familial cold auto inflammatory syndrome
MeSH Terms: conditions — Arthritis, Juvenile; Bronchiolitis Obliterans Syndrome; Arthralgia; Rheumatoid Arthritis, Systemic Juvenile; Mevalonate Kinase Deficiency; Cryopyrin-Associated Periodic Syndromes | interventions — canakinumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- canakinumab (Experimental): Patients will continue the same dose as their last dose administered in the study CACZ885G2301E1, CACZ885N2301 or CACZ885G2306. For all indications, the maximum canakinumab dose is 4 mg/kg or 300 mg for patients ≥ 40 kg. Ilaris® dosage may be adjusted (or interrupted) according to the clinical response and to investigators judgment.
  Interventions: Drug: canakinumab

INTERVENTIONS:
Drug: canakinumab — canakinumab

SUMMARY:
The objective of this extension protocol is to collect safety data (serious and non-serious adverse events) and to provide continuous canakinumab to patients in France who completed study CACZ885G2301E1(NCT00891046), CACZ885G2306 (NCT02296424) or CACZ885N2301 (NCT02059291) until a decision regarding reimbursement in France is effective for canakinumab (Ilaris®) in these indications.

ELIGIBILITY:
Inclusion Criteria

Criteria applicable for patients with Systemic Juvenil Idiopathic Arthritis SJIA):

Patients who have completed the international studies CACZ885G2301E1 or CACZ885G2306 without any significant safety issue according to Investigator's opinion.

Patients who have completed the international CACZ885G2306 study and who successfully withdrew canakinumab treatment per protocol but with a disease relapse after the end of study visit will be allowed to participate in CACZ885GFR01 study (whatever the time of relapse from the end of study visit), if the investigator states that there is an indication to resume canakinumab.

Patients who have participated in the international CACZ885G2306 study but could not be randomized and then have continued canakinumab in part I until the end of the study at a dose of 4 mg/kg every 4 weeks may be switched to CACZ885GFR01 study if the investigator thinks that, in the interest of the patient, there is an indication to taper off canakinumab dose after a prolonged remission.

Criteria applicable for patients with HPF (TRAPS, HIDS, crFMF):

Patients who have completed the international CACZ885N2301 study without any significant safety issue according to Investigator's opinion.

Criteria applicable for all patients:

Parent's or legal guardian's written informed consent and child's assent, if appropriate, or patient's written informed consent for patients ≥ 18 years of age must be obtained before any study related activity or assessment is performed.

Exclusion Criteria:

* History of recurring infections
* Hypersensitivity to the active substance or to any of the excipients

other protocol-defined inclusion/exclusion criteria may apply

Ages: 5 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 31 (Actual)
Dates: Start 2014-11-03 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2018-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (3):
- France (3):
  - Novartis Investigative Site, Bron
  - Novartis Investigative Site, Le Kremlin-Bicêtre
  - Novartis Investigative Site, Paris

IPD SHARING:
Plan to Share IPD: Undecided
Novartis is committed to sharing access to patient-level data and supporting clinical documents from eligible studies with qualified external researchers. Requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to protect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Canakinumab: Patients continued same dose as their last dose administered in the study CACZ885G2301E1, CACZ885N2301 or CACZ885G2306. For all indications, the maximum canakinumab dose was 4 mg/kg or 300 mg for patients ≥ 40 kg. Ilaris® dosage may have been adjusted (or interrupted) according to the clinical response and to investigator's judgment.
Period: Overall Study
Arm/Group | Canakinumab
Started (31) | 31
Completed (23) | 23
Not Completed | 8
Not completed — Adverse Event | 1
Not completed — Inclusion in the CACZ8852306 study | 1
Not completed — Patient no longer required study drug | 2
Not completed — Lack of Efficacy | 4

BASELINE CHARACTERISTICS:
Population: All patients
Arm/Group | Canakinumab
Number analyzed (Participants) | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.7 (4.07)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 14
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 29
  Other | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: The objective of this protocol was to collect additional safety data (serious and non serious AEs) and to provide continuous Ilaris® (canakinumab) treatment to patients in France who completed CACZ885G2301E1, CACZ885N2301 or CACZ885G2306 studies.
Time Frame: every 4 weeks up to 1 year
Population: Safety set: Safety set consisted of all patients who received at least one dose of study drug and had at least one post-treatment safety assessment in the study.
Measure: Count of Participants; unit: Participants
Groups:
- Canakinumab: Patients continued same dose as their last dose administered in the study CACZ885G2301E1, CACZ885N2301 or CACZ885G2306. For all indications, the maximum canakinumab dose is 4 mg/kg or 300 mg for patients ≥ 40 kg. Ilaris® dosage may have been adjusted (or interrupted) according to the clinical response and to investigators judgment.
Arm/Group | Canakinumab
Number analyzed (Participants) | 31
Participants
  Serious adverse events | 7
  Treatment emergent adverse events | 29

2. Primary Outcome: All-cause Mortality
Description: Number of participants who died for any reason during the study
Time Frame: uo to 1 year
Population: Safety set
Measure: Count of Participants; unit: Participants
Arm/Group | Canakinumab
Number analyzed (Participants) | 31
Participants | 0

ADVERSE EVENTS:
Time Frame: AEs and SAEs were collected for the maximum duration of treatment and follow up for a participant per protocol for approximately 12 months. All cause mortality (deaths) was collected from First Patient First Visit (FPFV) to Last Patient Last Visit (LPLV) up to a maximum of 1 year
Description: All cause mortality (deaths) was collected for as long as participants could be contacted from First Patient First Visit (FPFV) until Last Patient Last Visit (LPLV) up to a maximum of 1 year
Groups:
- Canakinumab (ACZ885): Patients continued the same dose as their last dose administered in the study CACZ885G2301E1, CACZ885N2301 or CACZ885G2306. For all indications, the maximum canakinumab dose is 4 mg/kg or 300 mg for patients ≥ 40 kg. Ilaris® dosage may have been adjusted (or interrupted) according to the clinical response and to investigators judgment.
Arm/Group | Canakinumab (ACZ885)
All-Cause Mortality (participants affected / at risk) | 0/31
Serious Adverse Events (participants affected / at risk) | 7/31
Other Adverse Events (participants affected / at risk) | 28/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Canakinumab (ACZ885) (N=31)
Histiocytosis haematophagic (Blood and lymphatic system disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 2
Epstein-Barr virus infection (Infections and infestations) | 1
Salmonellosis (Infections and infestations) | 1
Intentional overdose (Injury, poisoning and procedural complications) | 1
Scar (Injury, poisoning and procedural complications) | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 2
Bone disorder (Musculoskeletal and connective tissue disorders) | 1
Hallucination, auditory (Psychiatric disorders) | 1
Suicide attempt (Psychiatric disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Canakinumab (ACZ885) (N=31)
Lymphadenopathy (Blood and lymphatic system disorders) | 3
Abdominal pain (Gastrointestinal disorders) | 6
Abdominal pain upper (Gastrointestinal disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 4
Mouth ulceration (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 2
Toothache (Gastrointestinal disorders) | 2
Asthenia (General disorders) | 3
Pyrexia (General disorders) | 7
Bronchitis (Infections and infestations) | 3
Conjunctivitis (Infections and infestations) | 4
Gastroenteritis (Infections and infestations) | 7
Influenza (Infections and infestations) | 4
Labyrinthitis (Infections and infestations) | 2
Molluscum contagiosum (Infections and infestations) | 2
Nasopharyngitis (Infections and infestations) | 11
Onychomycosis (Infections and infestations) | 2
Oral herpes (Infections and infestations) | 2
Paronychia (Infections and infestations) | 4
Pharyngitis (Infections and infestations) | 4
Rhinitis (Infections and infestations) | 4
Sinusitis (Infections and infestations) | 2
Tonsillitis (Infections and infestations) | 4
Tracheitis (Infections and infestations) | 4
Viral infection (Infections and infestations) | 4
Ligament sprain (Injury, poisoning and procedural complications) | 2
Limb injury (Injury, poisoning and procedural complications) | 2
Iron deficiency (Metabolism and nutrition disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 9
Arthritis (Musculoskeletal and connective tissue disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 3
Juvenile idiopathic arthritis (Musculoskeletal and connective tissue disorders) | 3
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4
Pain in jaw (Musculoskeletal and connective tissue disorders) | 2
Scoliosis (Musculoskeletal and connective tissue disorders) | 2
Tendon pain (Musculoskeletal and connective tissue disorders) | 2
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Headache (Nervous system disorders) | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 2
Dry skin (Skin and subcutaneous tissue disorders) | 2
Eczema (Skin and subcutaneous tissue disorders) | 4
Rash (Skin and subcutaneous tissue disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2017-12-15): https://cdn.clinicaltrials.gov/large-docs/48/NCT02334748/Prot_000.pdf
  • Statistical Analysis Plan (2018-08-31): https://cdn.clinicaltrials.gov/large-docs/48/NCT02334748/SAP_001.pdf